CLINICAL TRIAL: NCT01655992
Title: A Randomized Open Label Multicenter Phase 3 Trial Comparing S1 Generic With Capecitabine in Patients With Metastatic Breast Cancer.
Brief Title: A Trial Comparing S1 Generic With Capecitabine in Metastatic Breast Cancer (MBC)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The sponsor decided to stop the study.
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, Vice Director of department of medical oncology, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fudan BR2012-09 CBCSG011
Record Dates: First submitted 2012-07-27; First posted 2012-08-02 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Metastatic Breast Cancer
Keywords: capecitabine; Tegafur，Gimeracil and Oteracil Potassium Capsules
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; potassium oxonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- S1 generic (Experimental): 40mg／m2 bid four weeks on two weeks off
  Interventions: Drug: S1 generic
- capecitabine (Active Comparator): 2500mg／m2／day divided into twice two weeks on one week off
  Interventions: Drug: capecitabine

INTERVENTIONS:
Drug: capecitabine — 2500mg／m2／day divided into twice two weeks on one week off
  Other Names: Xeloda
  Arms: capecitabine
Drug: S1 generic — 40mg／m2 bid four weeks on two weeks off
  Other Names: Tegafur，Gimeracil and Oteracil Potassium Capsules
  Arms: S1 generic

SUMMARY:
Comparing S1 generic With Capecitabine in Patients With Metastatic Breast Cancer.

DETAILED DESCRIPTION:
Comparing S1 generic(Tegafur，Gimeracil and Oteracil Potassium Capsules) With Capecitabine in Patients With Metastatic Breast Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast cancer
* Pretreated metastatic breast cancer not more than 2 lines chemotherapy
* Have not been previously treated with capecitabine,oral fluracil
* ECOG performance status of ≤ 1
* Be female and ≥ 18 and ≤ 75 years of age
* Have at least one target lesion according to the RECIST criteria 1.1

Exclusion Criteria:

* Pregnant or lactating women
* ECOG ≥ 2
* Have been treated with capecitabine
* Evidence of CNS metastasis
* History of another malignancy within the last five years except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix or a contralateral breast cancer
* Abnormal laboratory values: hemoglobin < 10.0 g/dl, absolute neutrophil count < 1.5×10^9/L, platelet count < 100×10^9/L, serum creatinine > upper limit of normal (ULN), serum bilirubin > ULN, ALT and AST > 5×ULN, AKP > 5×ULN
* Serious uncontrolled intercurrent infection
* Life expectancy of less than 3 months

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Estimated)
Dates: Start 2012-01; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
progression free survival | 6 months

SECONDARY OUTCOMES:
response rate | 1.5 months
overall survival | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Xi-chun Hu, MD,PhD, Principal Investigator — Fudan Univeristy Cancer Hospital
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China